CLINICAL TRIAL: NCT05746806
Title: A Single Arm Phase II Trial of Ultrahypofractionated Focal Salvage Radiotherapy for Isolated Prostate Bed Recurrence After Radical Prostatectomy
Brief Title: Trial of Ultrahypofractionated Focal Salvage Radiotherapy for Isolated Prostate Bed Recurrence After Radical Prostatectomy
Acronym: HypoFocal SRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Debiopharm International SA (Industry); Werner und Hedy Berger-Janser - Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01026
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Prostate Cancer
Keywords: Prostate; Salvage Radiation; Local recurrence; Stereotactic radiotherapy; Hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patients with locally recurred prostate cancer will receive a ultrahypofractionated stereotactic radiotherapy to the radiologically identified lesion (Dose: 5 fractions with 7Gray every second work week day) combined with an androgen deprivation therapy (LHRH-agonist / -antagonist) for 6 months.
  Interventions: Radiation: Ultrahypofractionated salvage radiotherapy to a local recurrence after radical prostatectomy; Drug: Androgen deprivation therapy

INTERVENTIONS:
Radiation: Ultrahypofractionated salvage radiotherapy to a local recurrence after radical prostatectomy — Ultrahypofractioned radiotherapy for patients with isolated local recurrence after radical prostatectomy in 5 fractions
Drug: Androgen deprivation therapy — In combination to the radiotherapy a short term androgen deprivation drug for 6 months will be applied.
  The preferred drug concept used is:
  - LHRH(Luteinizing hormone releasing hormone)-agonist with 3-month subcutaneous depot injection (e.g. Pamorelin® LA (Triptorelin) 11.25mg s.c.) in combination with nonsteroidal antiandrogen (e.g. Bicalutamide 50mg/day) as flare protection at least 5 days before and max. 15 days after first LHRH-injection
  Alternatively the following oral drug concept can be used, if the patient rejects injections:
  - GnRH (gonadotropin-releasing hormone)-antagonist with tablet intake for 6 months (e.g. Orgovyx® Tablets 120mg; first day 360mg, after second day 120mg per day)

SUMMARY:
The main objective of the trial is to explore the efficacy and safety of combining short-term androgen deprivation therapy (ADT) over 6 months to focal ultrahypofractionated salvage radiotherapy (SRT) delivered in 5 fractions to the site of local recurrence within the prostate bed after radical prostatectomy where multiparametric magnetic resonance imaging (mpMRI) and prostate-specific membrane antigen (PSMA) PET/CT are used to precisely identify the local recurrence and compare it to previously published literature.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent according to ICH/GCP (International Council for Harmonisation/Good Clinical Practice) regulations before registration and prior to any trial specific procedures
2. Age ≥ 18 years at time of registration
3. WHO performance status 0-1
4. Lymph node negative adenocarcinoma of the prostate treated with radical prostatectomy (RP) at least 6 months before trial.Tumor stage pT2a-3b, R0-1, pN0 or cN0. according to the Union for International Cancer Control (UICC) TNM 2009.
5. Evidence of measurable local recurrence at the prostate bed detected by PSMA PET/CT and mpMRI within the last 3 months. In case of unclear local recurrence, a biopsy confirmation is recommended.
6. Patient must have non-metastatic (N0, M0) disease, as defined by a lack of nodal or distant metastases seen on PSMA PET/CT scan
7. Patients must have non-castrate levels of serum testosterone (≥50 ng/dL).
8. Patients must not have previously received hormonal therapy (LHRH agonists, antiandrogen, or both, or bilateral orchiectomy).
9. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

1. Persistent PSA (> 0.4 ng/mL) 4 to 20 weeks after RP
2. Previous hematologic or primary solid malignancy within 3 years prior registration with the exception of curatively treated localized non-melanoma skin cancer
3. Usage of products known to affect PSA levels within 4 weeks prior to start of trial treatment phase including any form of androgen suppression agents and androgen deprivation therapy
4. Bilateral hip prosthesis
5. Severe or active co-morbidity likely to impact on the advisability of SRT
6. Treatment with any experimental drug or participation within a clinical trial within 30 days prior to registration (exception: concurrent participation in the biobank studies is allowed)

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical relapsefree survival | 2 years
  The initial prostate specific antigen (PSA) at time of registration will be the starting point. Freedom from biochemical progression is counted from the day of registration to the day of either first recorded biochemical progression as defined below, clinical progression or death due to clinical progression.
  Biochemical relapsefree survival measured with PSA (prostate specific antigen) lab testing at 1, 3, 6, 12, 18 and 24 months after radiotherapy. The duration of biochemical relapsefree survival is measured and documented in months for each patient.
  A biochemical recurrence is defined by any confirmed PSA rise above 0.20 ng/mL with a confirmatory rise at least 2 weeks later. For those patients whose PSA does not drop below 0.20 ng/mL at time of first response assessment at 3 months are considered as non-responders to treatment and are considered to have a biochemical recurrence in case a second measurement at least 2 weeks later confirms a rising PSA above this level.

SECONDARY OUTCOMES:
Acute side effects of grade 3 or higher | 90 days
  Standard acquisition of therapy related acute side effects of grade 3 or higher according to NCI CTCAE v5.0 at radiotherapy end and at 1 and 3 months after radiotherapy will be assessed. The side effects are recorded with the corresponding grade according to the NCI CTCAE v5.0 scale at the measured points of time.
  Special attention shall be given to diarrhea, fecal incontinence, proctitis, rectal hemorrhage, rectal pain, hematuria, urinary frequency, urinary urgency, urinary retention, urinary incontinence, cystitis non-infective and erectile dysfunction.
Clinical progression-free survival | 2 years
  Clinical progression-free survival is defined as time between registration and the appearance of a new recurrence (any N1 or M1) as suggested by PET-CT, symptoms related to progressive prostate cancer (PC), or death due to any cause.
  The duration of clinical progression-free survival is measured and documented in months for each patient.
  Definition of recurrence:
  * A local recurrence is defined as the appearance of evidence of a recurrence within the prostate bed. Confirmation of the recurrence by biopsy is recommended, whenever possible.
  * A regional nodal recurrence is defined as a radiographic (PET-CT) evidence of a lymphadenopathy in the pelvis in a patient without the diagnosis of hematologic/lymphatic disorder
  * Distant recurrence is defined as the appearance of distant metastases (M1a, M1b, M1c) outside the pelvis.
Metastasis-free survival | 2 years
  Metastasis-free survival is defined as time between registration and the appearance of a metastatic recurrence (any M1) as suggested by PET-CT or death due to any cause. The duration of metastasis-free survival is measured and documented in months for each patient.
  Patients without any of the events of interest (including those with biochemical relapse only) are censored at the date of the last follow-up. Second cancers are not considered events in terms of this endpoint. In case of biochemical progression, re-staging will be made with PET-CT imaging preferably with the same tracer used before registration. In case of negative PET findings at biochemical relapse, a new PET imaging should be repeated on a 6-monthly basis or earlier in case clinically indicated.
Late side effects | After 90 days up to 2 years (after acute side effects, see outcome 2)
  Standard acquisition of therapy related late side effects according to NCI CTCAE v5.0 at 6, 12, 18 and 24 months after radiotherapy. The side effects are recorded with the corresponding grade according to the NCI CTCAE v5.0 scale at the measured points of time.
  Special attention shall be given to diarrhea, fecal incontinence, proctitis, rectal hemorrhage, rectal pain, hematuria, urinary frequency, urinary urgency, urinary retention, urinary incontinence, cystitis non-infective and erectile dysfunction.
Quality of life (EORTC Quality of life questionnaire C-30 version 3) | 2 years
  All patients registered into this trial are to complete QoL questionnaires at registration and at 1, 3, 6, 12, 18, 24 months after radiotherapy. A longitudinal design is used. Patients are asked to complete the EORTC Quality of life questionnaire C-30 version 3. The resulting score will be documented at each point of time.
Quality of life ( EORTC Quality of life PR25) | 2 years
  All patients registered into this trial are to complete QoL questionnaires at registration and at 1, 3, 6, 12, 18, 24 months after radiotherapy. A longitudinal design is used. Patients are asked to complete the EORTC Quality of life questionnaire PR25 prostate cancer module. The resulting score will be documented at each point of time.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MS Shelan, PD, Study Director — Department of radiation oncology, Bern University Hospital, Inselspital, Berne, Switzerland
Locations (5):
- Switzerland (5):
  - Universitätsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana-Ente Ospedaliero Cantonale (IOSI-EOC), Bellinzona
  - Inselgruppe AG, Inselspital, Bern
  - Kantonsspital Winterthur, Klinik für Radio-Onkologie, Winterthur
  - Universitätsspital Zürich, Klinik für Radio-Onkologie, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathier E, Althaus A, Zwahlen D, Lustenberger J, Zamboglou C, De Bari B, Aebersold DM, Guckenberger M, Zilli T, Shelan M. HypoFocal SRT Trial: Ultra-hypofractionated focal salvage radiotherapy for isolated prostate bed recurrence after radical prostatectomy; single-arm phase II study; clinical trial protocol. BMJ Open. 2024 Jan 30;14(1):e075846. doi: 10.1136/bmjopen-2023-075846. PMID 38296279

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT05746806/Prot_SAP_002.pdf